CLINICAL TRIAL: NCT05380167
Title: Efficacy and Variability in Plasma Nitrite Levels During Long-term Supplementation With Nitrate Containing Beetroot Juice
Brief Title: Efficacy Long-term Dietary Nitrate Consumption to Plasma Nitrite Conversion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Principal Investigator, Gary Miller, Professor, Wake Forest University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB000022922
Record Dates: First submitted 2022-05-12; First posted 2022-05-18 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Cardiovascular Diseases in Old Age
Keywords: beetroot juice; dietary nitrate; plasma nitrite

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into one of two groups. The first group will consume daily beetroot juice containing 380 mg of nitrate and the second group will consume daily beetroot juice with nitrate removed.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A third party not involved with the conduct of the study provided research staff with the beetroot juice in participant specific coded bottles. The research staff then distributed these coded bottles to the participant. At the end of the trial, the code was revealed for intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BRJ Nitrate (Experimental): This arm consumed daily for 12 weeks a 70 mL bottle of beetroot juice containing 380 mg of nitrate.
  Interventions: Dietary Supplement: BRJ Nitrate
- BRJ Placebo (Placebo Comparator): This arm consumed daily for 12 weeks a 70 mL bottle of beetroot juice containing 0 mg of nitrate.
  Interventions: Dietary Supplement: BRJ Placebo

INTERVENTIONS:
Dietary Supplement: BRJ Nitrate — Participants in this group drank daily for 12 weeks a 70 mL bottle of Beet It Sport drink with nitrate.
  Arms: BRJ Nitrate
Dietary Supplement: BRJ Placebo — Participants in this group drank daily for 12 weeks a 70 mL bottle of Beet It Sport drink without nitrate
  Arms: BRJ Placebo

SUMMARY:
The objective of this study was to determine the chronic effects of beetroot juice supplementation on the acute (90-minute post nitrate consumption) efficacy of converting dietary nitrate to plasma nitrate and plasma nitrite in healthy middle-to-older aged adults. the investigators were also interested in determining the effect of this intervention on fasting levels of plasma nitrate and nitrite over time. Furthermore, the number of participants classified as "non-responders" was determined based on increases in plasma nitrite achieved using tolerable volumes of beetroot juice by other studies.

ELIGIBILITY:
Inclusion Criteria:

* Middle and Older (40-80 year-old) men and women
* Body mass index between 18.5 - 30.0 kg/m2
* Able to provide own transportation to study testing visits
* Able to consume study beverages
* Able to speak and read English

Exclusion Criteria:

* Tobacco user (smoke or chew), including e-cigarettes
* Known conditions of: diabetes mellitus (type 1 or 2), atrophic gastritis, hypo- or hyperthyroidism, gout, history of kidney stones, history of hypotension, cardiovascular disease, chronic obstructive pulmonary disease, inflammatory bowel diseases, impaired liver or kidney function
* Current or recent (last 3 months) treatment for cancer
* Current use of the following medications: Phosphodiesterase type 5 inhibitors, nitroglycerin or nitrate preparations, proton pump inhibitors, medication for hypothyroidism, antacid and heartburn medications

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Fasting Plasma Nitrate | Collected at baseline (week 0), end of week 1, week 2, week 3, week 4, week 8, and week 12
  Concentration of nitrate in the plasma obtained at the start of each testing visit
Fasting Plasma Nitrite | Collected at baseline (week 0), end of week 1, week 2, week 3, week 4, week 8, and week 12
  Concentration of nitrite in the plasma obtained at the start of each testing visit
90 minute plasma Nitrate | Collected at baseline (week 0), end of week 1, week 2, week 3, week 4, week 8, and week 12
  Concentration of nitrate in the plasma obtained 90 minutes following the consumption of the intervention arm's assigned beverage
90 minute plasma Nitrite | Collected at baseline (week 0), end of week 1, week 2, week 3, week 4, week 8, and week 12
  Concentration of nitrite in the plasma obtained 90 minutes following the consumption of the intervention arm's assigned beverage

CONTACTS AND LOCATIONS:
Locations (1):
- Wake Forest University, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No